CLINICAL TRIAL: NCT02615964
Title: 'Defining the Gold Standard in Diagnosis and Stratification of Raynaud's Disorder', Nova Cold Hands Raynaud's Disorder. Raynaud's Disease is a Vascular Disorder Which Results in Decreased Blood Flow to the Hands and Feet.
Brief Title: Nova Cold Hands Raynaud's Disorder, a Disease Which Results in Decreased Blood Flow to the Hands and Feet.
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Nadera J. Sweiss, Associate Professor of Medicine, University of Illinois at Chicago
Other Study IDs: 2014-1128
Record Dates: First submitted 2015-07-08; First posted 2015-11-26 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Raynaud's Disease
MeSH Terms: conditions — Raynaud Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Nova Flow Procedure — Evaluation of the diagnosis, and stratification of the severity of Raynaud's disorder in patients with scleroderma based on clinical and imaging data will allow creation of more precise diagnostic criteria as well as disease classification which may guide treatment practices. The study results will likely have no immediate benefit to the patients participating in the study, however may have a future impact diagnosis, stratification and ultimately treatment of patients with Raynaud's disorder. In addition, data collected in this study may provide insight into disease process and leading to future research endeavors.

SUMMARY:
Patients presenting to UIC rheumatology clinic with Raynaud's disorder and scleroderma will be asked to participate. 10 hands of patients with both Raynaud's disorder and scleroderma will be studied. This research study is being done to better understand Raynaud's disease and to assess the role of blood flow measurement in diagnosing the disorder, specifically, through data collected by an MRI procedure called NOVA FLOW. NOVA is a blood flow measurement software system owned by the study's sponsor, VasSol, Inc.

DETAILED DESCRIPTION:
The investigators propose to obtain volumetric flow data on 10 hands of patients with Raynaud's disorder and scleroderma at UIC rheumatology clinic and compare these results with previously established volumetric flow data for non-Raynaud's patients. Through this analysis, the invstigators will be able to better understand and correlate subjective and objective measures of both disease presentation and progression. Collection of cross sectional data will allow us to better address the following questions Is it possible to more precisely diagnose patients with Raynaud's disorder based on NOVA analysis as well as clinical findings

Is it possible to stratify patients with Raynaud's disorder into categories which may allow:

i. Prediction of disease course and prognosis ii. Prediction of response to specific treatment modalities (vasodilators vs anti-coagulation vs surgical or chemical denervation) The investigators propose to collect measurements of disease severity as well as functional assessment of patients Raynaud's and scleroderma in order to address the following questions c. Does NOVA flow and volume data correlate with measures of Raynaud's and scleroderma disease severity index d. Does NOVA flow and volume data correlate with OT assessment of hand functionality.

ELIGIBILITY:
Inclusion Criteria:

* Inclusionary criteria for this study will be patients with a diagnosis of Raynaud's disease and scleroderma (per ACR criteria for the diagnosis for systemic sclerosis) and age between 18-85.

Exclusion Criteria:

* Exclusion criteria for Raynaud's patients will include history of botox injection to the hands within 6 months, non-English speaking patients and those unable to understand informed consent, and the presence of confounding medical conditions preventing the patient from full participation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to UIC rheumatology clinic with Raynaud's disorder and scleroderma will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The measurement of blood flow | Up to one year
  There will be two visits in the study. Each of those visits will take about one hour.
  * First visit will consist of: NOVA flow procedure, Medical history, Digital photographic assessments, Nail bed capillaroscopy and questionnaires.
  * Second visit will occur one month after the first visit and consist of: Follow up for any adverse events due to the study. Review any changes with the hands that received the NOVA procedure. Complete any follow up questionnaires needed for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nadera J Sweiss, MD, Principal Investigator — University of Illinois at Chicago